CLINICAL TRIAL: NCT01947517
Title: The Retention Rate Between Superflex Punctal Plugs, and Parasol Punctal Occluders
Brief Title: The Retention Rate Between Brand A and Brand B Punctal Plugs
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephanie Baxter, Program Director Department of Ophthalmology, Queen's University
Other Study IDs: Punctal plugs
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parasol Punctal Occluder Group: Randomized to receive Brand A punctal plugs
  Interventions: Device: Parasol Punctal Occluder
- Superflex Punctal Occluder Group: Randomized to receive Group B punctal plugs
  Interventions: Device: Superflex Punctal Occluder

INTERVENTIONS:
Device: Parasol Punctal Occluder — Patients will be randomized to receive one of these 2 punctal occluders in the management of dry eyes.
  Groups: Parasol Punctal Occluder Group
Device: Superflex Punctal Occluder — Patients will be randomized to receive one of these 2 punctal occluders in the management of dry eyes.
  Groups: Superflex Punctal Occluder Group

SUMMARY:
The purpose of this study is to determine if Parasol punctal occluders (Brand A) have a higher rate of retention than Superflex punctal plugs (Brand B).

DETAILED DESCRIPTION:
Eyes will be randomized to either Brand A or Brand B punctal plug. The primary outcome measure is length of time punctual plugs are retained, measured in months. This will be measured at monthly assessments for 6 months. Secondary outcome measures include patient satisfaction, and improvement in subjective and objective dry eye scores, as well as complications related to punctual plugs including spontaneous plug loss, and intolerance. We will evaluate these measures by repeating the Canadian Dry Eye Assessment, Schirmer 1, tear meniscus height, fluorescein corneal staining (NEI scale), and lissamine green conjunctival staining (NEI scale) at month 1, month 3, and month 6 visits.

ELIGIBILITY:
Inclusion Criteria:

* moderate dry eye, severe dry eye

Exclusion Criteria:

* silicone allergy, punctal stenosis, punctal occlusion, punctal cautery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from cornea and general ophthalmology specialist practices at Hotel Dieu Hospital, Queens University
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley R Brissette, BSc, MD, Study Director — Queens University; Stephanie Baxter, MD, FRCSC, Principal Investigator — Queens University
Locations (1):
- Department of Ophthalmology, Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Parasol Group: Randomized to receive Brand A punctal plugs
  Parasol Punctal Occluder
- Superflex Group: Randomized to receive Group B punctal plugs
  Superflex Punctal Occluder
Period: Overall Study
Arm/Group | Parasol Group | Superflex Group
Started | 26 | 26
Completed | 25 | 25
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parasol Group | Superflex Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (17.67) | 58.4 (16.18) | 60.1 (15.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Length of Retention
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Parasol Group | Superflex Group
Number analyzed (Participants) | 25 | 25
months | 6 (0) | 6 (0)

2. Secondary Outcome: Canadian Dry Eye Assessment Score
Description: Describes the scores on a scale and range from 0-3. Higher score represents more severe dry eye. Score 0 = no dry eye symptoms, score 1 = mild dry eye symptoms, score 2 = moderate dry eye symptoms, score 3 = severe dry eye symptoms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parasol Group | Superflex Group
Number analyzed (Participants) | 25 | 25
scores on a scale | 1.06 (1.081) | 0.25 (1.018)

3. Secondary Outcome: National Eye Institute Corneal Fluorescein Staining Pattern
Description: The cornea is divided into 5 zones, and the inferior zone 5 was assessed for staining pattern. Grade 0= no staining, grade 1= trace staining, grade 2= mild staining, grade 3= moderate staining, and grade 4= severe staining.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Parasol Group | Superflex Group
Number analyzed (Participants) | 25 | 25
Scores on a scale | 3.28 (1.091) | 3.60 (0.756)

4. Secondary Outcome: National Eye Institute Grading for Conjunctival Staining
Description: The conjunctival staining is divided into 6 zones. Each zone received a score for staining with lissamine green. Grade 0= no staining, grade 1= trace staining, grade 2= mild staining, grade 3= moderate staining, grade 4= severe staining. Data from different zones was combined and the total value was averaged.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Parasol Group | Superflex Group
Number analyzed (Participants) | 25 | 25
Scores on a scale | 2.08 (0.895) | 2.08 (0.463)

5. Secondary Outcome: Tear Meniscus Height
Description: Meniscus height measured in mm
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Parasol Group | Superflex Group
Number analyzed (Participants) | 25 | 25
mm | 0.472 (0.398) | 0.468 (0.217)

ADVERSE EVENTS:
Arm/Group | Parasol Group | Superflex Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No